CLINICAL TRIAL: NCT06824896
Title: An Observational Database Study to Monitor Safety-related Endpoints After Marketing of Cecolin®
Brief Title: A Post-marketing Observational Database Study Monitoring the Safety of CecolinⓇ
Acronym: HPV-PRO-013
Status: Completed | Type: Observational
Sponsor: Xiamen Innovax Biotech Co., Ltd (Industry)
Collaborators: Xiamen University (Other); Xiamen Health and Medical Big Data Center (Unknown)
Responsible Party: Sponsor
Other Study IDs: HPV-PRO-013
Record Dates: First submitted 2025-01-24; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Autoimmune Diseases; Adverse Pregnancy Outcomes
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- premarketing corhort: females aged 9-45 years during premarketing observation of CecolinⓇ
- postmarketing corhort: females aged 9-45 years during postmarketing observation of CecolinⓇ

SUMMARY:
This study was a retrospective-prospective real-world study to assess the safety among females receiving the 2vHPV vaccine (CecolinⓇ).

DETAILED DESCRIPTION:
This study was initiated following the approval of the Recombinant Human Papillomavirus Bivalent (Types 16, 18) Vaccine (Escherichia coli) (CecolinⓇ) in China. We undertook a retrospective-prospective real-world study to assess the incidence of new-onset autoimmune conditions (10 conditions in rheumatologic/hematologic, gastroenterologic, endocrinologic, and ophthalmologic) and adverse pregnancy conditions (e.g., premature birth, birth defects) among 9-45 yoa females during the pre- and post-marketing period of CecolinⓇ.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 9 to 45 years registered at the Xiamen Health and Medical Big Data Center;
* Having at least two records in the Xiamen Health and Medical Big Data Center with an interval of 12 months or more.

Exclusion Criteria:

-

Ages: 9 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: * Females aged 9 to 45 years registered at the Xiamen Health and Medical Big Data Center;
  * Having at least two records in the Xiamen Health and Medical Big Data Center with an interval of 12 months or more.
Sampling Method: Non-Probability Sample
Enrollment: 1322084 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
autoimmune conditions | through study completion, around 7.3 years
  incidence of autoimmune conditions in rheumatologic/hematologic, gastroenterologic, endocrinologic, and ophthalmologic
adverse pregnancy conditions | through study completion, around 7.8 years
  incidence of the adverse pregnancy outcomes in maternal, fetal and neonatal

SECONDARY OUTCOMES:
other serious diseases | through study completion, around 7.3 years
  incidence of primary ovarian insufficiency, facial paralysis, complex regional pain syndrome and postural orthostatic tachycardia syndrome.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiamen Innovax Biotech Co., Ltd, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No